CLINICAL TRIAL: NCT07155551
Title: Measuring Changes In Choroidal Thickness Induced By Prototype Soft Contact Lenses Worn For 1 Hour
Acronym: ARCTIC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Myoptechs, Inc (Industry)
Collaborators: University of Waterloo School of Optometry and Vision Science (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Other
Other Study IDs: P/883/24/MO
Record Dates: First submitted 2025-08-15; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Myopia; Refractive Error
MeSH Terms: conditions — Myopia; Refractive Errors

STUDY DESIGN:
Intervention Model Description: We understand that this falls outside the realm of a feasibility study given the intended sample size of 20 subjects. That being stated we selected Other in our resubmission, because in our opinion none of the "Primary Purpose" selection options fit the intent of studying the contact lenses impact on the choroid to detect the eyes' ability to respond to the defocus created by these lenses. These data will help inform further development decisions for an eventual clinical trial.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (3):
- Lens A (Experimental)
  Interventions: Device: Lens A; Device: Lens B; Device: Lens C
- Lens B (Experimental)
  Interventions: Device: Lens A; Device: Lens B; Device: Lens C
- Lens C (Experimental)
  Interventions: Device: Lens A; Device: Lens B; Device: Lens C

INTERVENTIONS:
Device: Lens A — Lens A of Study P/883/24/MO
Device: Lens B — Lens B of Study P/883/24/MO
Device: Lens C — Lens C of Study P/883/24/MO

SUMMARY:
The objective of the study is to evaluate the short-term change in choroidal thickness induced by 3 prototype soft contact lenses for people with myopia.

ELIGIBILITY:
Inclusion Criteria:

* Are 18-25 years of age (inclusive) and have full legal capacity to volunteer; Have read (or be read to) and signed the information and consent form; Habitually wear soft contact lenses or are spectacle wearers with previous experience of soft contact lens wear;
* Are myopic with both eyes having a vertex corrected spherical equivalent non-cycloplegic refraction of at least -0.50 DS and no more than -4.50 DS;
* Achieve at least LogMAR +0.10 with spherical equivalent refraction in each eye;
* Are willing and able to maintain the appointment schedule and follow the measurement visit instructions which include no use of caffeine drinks, alcohol or other stimulants 12 hours before each measurement visit and no smoking or use of recreational cannabis 24 hours before the study visit;
* Have not used a myopia control treatment within 2 years prior to Visit 0 (this includes multifocal spectacle or contact lens wear, orthokeratology, or atropine);
* Typically sleeps at least 7 hours per night.

Exclusion Criteria:

* Participating in any concurrent clinical or research study;
* Have astigmatism of more than 1.00 DC in either eye as per non-cycloplegic refraction;
* Have amblyopia in either eye or known to have any other binocular vision disorder, such as accommodative insufficiency;
* Have any known active* ocular disease and/or infection;
* Have a systemic condition that in the opinion of the investigator may affect a study outcome variable. Examples include diabetes mellitus, hyperthyroidism, and active allergies;
* Are using any systemic or topical medications that in the opinion of the investigator may affect a study outcome variable. Examples include antihistamine, atropine eye drops;
* Have known sensitivity to the sodium fluorescein diagnostic pharmaceutical to be used in the study;
* Self-reports as pregnant, lactating or planning a pregnancy at the time of enrolment;
* Have undergone strabismus surgery, refractive error surgery or intraocular surgery;
* Are an employee of the Centre for Ocular Research & Education directly involved in this study (i.e. on the delegation log).

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-08-25 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in Choroidal Thickness from Baseline to After 1 Hour of Contact Lens Wear | After 1 hour of wearing each contact lens
  The change in sub-foveal choroidal thickness for the 3 study contact lenses will be compared from baseline to after 1 hour of contact lens wear. Measurements will be conducted on the right eye using a swept-source Optical Coherence Tomographer and measured in micrometers.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Ocular Research and Education at the School of Optometry and Vision Science at Waterloo University, Waterloo, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
The results are regarded as confidential to our business as Sponsor, and confidential for the selection of one device to use in a future efficacy trial. There are no plans for a public data repository for this study.